CLINICAL TRIAL: NCT06247904
Title: Noninvasive Brain Stimulation Therapy in Subacute Human Spinal Cord Injury: A Translational Study
Brief Title: NIBS Therapy in Subacute Spinal Cord Injury
Acronym: NIBS-SCI1
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Pennsylvania Department of Health (Other Government); University of Mississippi Medical Center (Other); University of Sao Paulo (Other); Massachusetts General Hospital (Other); Weill Medical College of Cornell University (Other); Burke Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dylan Edwards, Director, Jefferson Moss Rehabilitation Research Institute, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: iRISID-2023-2494
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Spinal Cord Injury; Tetraplegia/Tetraparesis
Keywords: Spinal cord injury; Cervical spinal cord; Transcranial Magnetic Stimulation; Recovery; Motor cortex
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be equally randomized to either the Active rTMS or Sham rTMS group following the Baseline Assessment. Device will be set up to active/sham mode prior to intervention using a unique patient and intervention code by an unblinded study team member. Subjects, outcome assessors and staff administering rTMS intervention (care provider) will be blinded to the device setting (Active/Sham).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): 10 daily sessions of High-frequency Transcranial Magnetic Stimulation (HF-rTMS) applied bilaterally over the hand primary motor area informed by e-field modelling and targeting will be aided by neuronavigation system for precise targeting during each intervention session. Active group will receive HF-rTMS intensity calculated using electric field modelling to create electric field intensity of approximately motor threshold, using the cool-B65 A/P rTMS coil.
  Interventions: Device: Active rTMS
- Sham rTMS (Sham Comparator): 10 daily sessions of Sham High-frequency Transcranial Magnetic Stimulation (HF-rTMS) applied bilaterally over the hand primary motor area informed by e-field modelling and targeting will be aided by neuronavigational system for precise targeting during each intervention session Sham group receives no active magnetic stimulation. Cool-B65 A/P rTMS coil will be used to avoid unblinding of administrator and/or study participant.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: Active rTMS — The stimulation protocol will comprise 15Hz pulse trains, each 50 pulses, repeated 10x, with a 60s inter-train interval. Stimulation intensity will be determined from individual MRI-modeled e-field, to achieve approximately motor threshold in the target area.
  Other Names: active repetitive transcranial magnetic stimulation
  Arms: Active rTMS
Device: sham rTMS — The stimulation protocol will comprise 15Hz pulse trains, each 50 pulses, repeated 10x, with a 60s inter-train interval. Stimulation intensity will be close to zero (negligible) since sham coil will be used for the intervention
  Other Names: sham repetitive transcranial magnetic stimulation
  Arms: Sham rTMS

SUMMARY:
No accepted clinical therapies exist for repair of motor pathways following spinal cord injury (SCI) in humans, leaving permanent disability and devastating personal and socioeconomic cost. A robust neural repair strategy has been demonstrated in preclinical studies, that is ready for translation to recovery of hand and arm function in human SCI, comprising daily transcranial magnetic stimulation treatment at the inpatient rehabilitation facility. This study will establish clinical effect size of the intervention, as well as safety and feasibility necessary for a subsequent controlled efficacy trial and inform preclinical studies for dosing optimization.

DETAILED DESCRIPTION:
The objective of this proposal is to begin translating findings from pre-clinical studies to human motor deficits following cervical SCI (cervSCI). This HF-rTMS treatment protocol has not been previously assessed in human SCI and is qualitatively different from rTMS protocols reported to transiently modulate excitability of existing pathways, previously demonstrated in the literature. The protocol involves a daily stimulation of ~10 mins bilateral HF-rTMS for 2 weeks. SCI participants will be studied in a United States inpatient setting for this phase I study.

Given the findings in the pre-clinical model of robust axonal sprouting and functional synapse formation close to the damaged tissue using the above stimulation parameters, the transcranial magnetic stimulation treatment will target the hand-forearm region of the primary motor cortex, bilaterally. The aim is to include the cortical representation of affected muscles adjacent to the neurological level of injury. This zone often contains a mix of clinically and neurophysiologically intact, weakly innervated and denervated corticospinal pathways. Under standard sub-acute rehabilitation care, recovery of up to 1 neurological level of injury (NLI) is often the case, but improvement of 2 or more levels is far less common (<30% of patients). To examine the feasibility and safety of this novel intervention is the principal aim of the study. The associated potential clinical and neurophysiological changes will also be evaluated. These preliminary data will be used to power a subsequent efficacy trial to test the hypothesis that rTMS induced corticospinal augmentation will result in greater than typical extension of the NLI in human SCI, assessed up to the stable recovery phase at 6 months post-injury.

ELIGIBILITY:
Inclusion Criteria:

1. Post traumatic or non-traumatic cervical spinal cord injury (SCI) with residual upper-extremity paralysis
2. Time post-injury less than six weeks
3. Neurological Level of Injury (NLI) C4-C6
4. ASIA Impairment Scale (AIS) A-D
5. Sensory and motor zone of partial preservation (ZPP, clinically complete or incomplete)
6. Age 18 to 80 years old

Exclusion Criteria:

1. Ventilator dependence;
2. Concurrent neurological condition affecting sensory or motor pathways or otherwise limiting ability to participate in the study;
3. Evidence of trauma-related brain injury;
4. Contraindications for TMS or history of seizure or seizure risk;
5. Spinal instability;
6. Uncontrolled autonomic dysreflexia;
7. Severe muscular or skeletal or neuropathic pain;
8. Known or suspected pregnancy;
9. Medically unstable or any reason the physician may deem as inappropriate for the participant to enroll or continue in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Eligibility - (Percentage candidates eligible of screened patients) | 21 months (Recruitment period)
  The proportion of patients who can take part in the study, whether they later agree to or not.
Recruitment - (Percentage candidates enrolled of approached patients) | 21 months (Recruitment period)
  The proportion of eligible patients who agree to take part in the study.
Adherence to intervention - (Percentage candidates who dropout during the intervention period of enrolled candidates) | 2 years (Duration of human subjects' involvement)
  Proportion of intervention-related dropouts.
Adherence to outcome assessment - (Percentage candidates who do not complete outcome assessments of enrolled candidates) | 2 years (Duration of human subjects' involvement)
  Proportion of patients that complete the assessments at the start and the end of the intervention.
Retention - (Percentage candidates who do not complete 6-month follow up of enrolled candidates) | 2 years (Duration of human subjects' involvement)
  The number of patients who drop out or were 'lost' at the 6-month follow-up.
Adverse Events | 2 years (Duration of human subjects' involvement)
  Rate of adverse and serious adverse events

SECONDARY OUTCOMES:
Motor neurological level change (ISNCSCI assessment) | Baseline and 6 months after injury
  Proportion of patients with Improvement of 2 or more motor zone of partial preservation levels from baseline to 6 months after injury.
Incidence of reconnectivity (Proportion: MEP absent, covert to MEP present) | Baseline and 6 months after injury
  The proportion of re-connectivity will be estimated by treatment group.
Change in motor threshold between groups (Difference in %Maximum Stimulator Output to achieve motor threshold) | Baseline and 6 months after injury
  Change in motor threshold of key muscles will be estimated bilaterally within each group and a comparison of the change between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan J Edwards, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Jefferson Moss-Magee Rehabilitation - Elkins Park, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, data will be deidentified and shared within the supplementary material of published scientific papers or per the journal recommendations. We may also share the full range of available individual participant data with the members of the scientific community upon reasonable request and at the discretion of the PI.
Supporting Information: SAP, Analytic Code
Time Frame: Data will become available upon publication of results and may be shared indefinitely.
Access Criteria: IPD and any additional supporting information will be shared with members of the scientific and medical communities for analyses related to the use of rTMS to improve upper extremity motor function following neurological insult. The mechanism for data sharing will be decided on a case by case basis; the study PI will review all data sharing request.